CLINICAL TRIAL: NCT03322917
Title: A Prospective Interventional Non-randomized and Non-comparative Series of Cases of Patiens Suffering Ocular Surface Syndrome Post-LASIK: Outcomes After the Treatment With Platelet Rich Plasma
Brief Title: Ocular Surface Syndrome Post-lasik, Outcomes of Treatment With Platelet Rich Plasma
Acronym: PRP-OSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vissum, Instituto Oftalmológico de Alicante (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRP-autologous/0208
Record Dates: First submitted 2017-10-18; First posted 2017-10-26 (Actual); Last update posted 2017-12-04 (Actual); Status verified 2017-12

CONDITIONS: Dry Eye After LASIK-Laser in Situ Keratomileusis
Keywords: dry eye; PRP; autologous; after LASIK; ocular surface
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Prospective interventional non-comparative consecutive case series.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: PRP autologous — Autologous platelet rich plasma: 1 drop / 6 times a day during 6 weeks

SUMMARY:
To evaluate the efficacy of autologous platelet-rich plasma eye drops (E-PRP) for the treatment of chronic ocular surface syndrome (OSS) following laser in situ keratomileusis (LASIK).

DETAILED DESCRIPTION:
Prospective interventional consecutive case series including 156 eyes of 80 patients affected by chronic post-LASIK OSS who were treated with autologous E-PRP 6 times a day as monotherapy for 6 weeks. Assessment after treatment with E-PRP included: dry eye symptoms, change in corrected distance visual acuity (CDVA), corneal fluorescein staining (CFS) and conjunctival hyperemia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients suffering from moderate to severe dry eye syndrome for 6 months or more after conventional treatments with artificial tears following LASIK.
* Tear break-up time (TBUT) between 4 and 9 seconds.

Exclusion Criteria:

* Ocular pathology needing topical treatments different than dry eye syndrome
* Trombocitopeny, associated pathologies to coagulation factors or any state of plaquets antiagregation (AAS and other AINES).
* Ocular tumours, corneal distrophies, history of ocular herpes.
* Pregnant or nursering women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-07-01 (Actual); Primary Completion 2013-01-17 (Actual); Study Completion 2013-01-17 (Actual)

PRIMARY OUTCOMES:
Corneal fluorescein staining (CFS) | Before LASIK surgery and after the 6 weeks of treatment
  Staining using fluorescein will be graded using the modified Oxford scale (7-point ordinal scale, score 0, 0.5, and 1 to 5 (see Appendix 2). On this modified scale, the score 0 corresponds to no staining dots and the score 0.5 to three or less staining dots. A CFS grade of 0 represents complete corneal clearing.
  A negative change from baseline will indicate improvement.

SECONDARY OUTCOMES:
Dry eye symptoms | Before LASIK surgery and after the 6 weeks of treatment
  The symptoms of ocular discomfort (unrelated to instillation of the study medication), burning/stinging, foreign body sensation, eye dryness, pain, will be assessed for intensity by the study patients using a self-administered VAS ranging from 0% to 100%. The symptoms will be assessed separately for each eye and data from the worst eye will be used for analysis.
  A decrease in the VAS score from baseline will indicate improvement.
Corrected distance visual acuity (CDVA) | Before LASIK surgery and after the 6 weeks of treatment
  Best corrected distance visual acuity (BCDVA) will be measured using the LogMar scale. The patient is seated at 3 or 4 m from the EDTRS or modified EDTRS chart, depending on chart size and must try to read all letters first while covering the left eye, then while covering the right eye.
Conjunctival hyperemia | Before LASIK surgery and after the 6 weeks of treatment
  Biomicroscopy will be performed using a slit lamp. The patient will be seated while being examined grading of the conjunctival hyperemia, according to the following scales:
  0 = None (normal).
  1. = Mild (a flush reddish color predominantly confined to the palpebral or bulbar conjunctiva).
  2. = Moderate (more prominent red color of the palpebral or bulbar conjunctiva).
  3. = Severe (definite redness of palpebral or bulbar conjunctiva).

CONTACTS AND LOCATIONS:
Overall Officials: JORGE L ALIO, DR., Principal Investigator — Vissum, Instituto Oftalmológico de Alicante

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alio JL, Rodriguez AE, Abdelghany AA, Oliveira RF. Autologous Platelet-Rich Plasma Eye Drops for the Treatment of Post-LASIK Chronic Ocular Surface Syndrome. J Ophthalmol. 2017;2017:2457620. doi: 10.1155/2017/2457620. Epub 2017 Dec 12. PMID 29379652